CLINICAL TRIAL: NCT05859204
Title: Impact of Exercise Groups on Patient Mental Health and Wellbeing in an Acute Psychiatric Inpatient Unit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00373975
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Hospitalization; Physical Inactivity; Depression, Anxiety; Sleep
MeSH Terms: conditions — Sedentary Behavior; Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT-led Exercise Group on Inpatient Psychiatry Unit (Experimental): Occupational therapist (OT) led group. Group includes education, warm-up, high intensity interval training cardio, strength, kick boxing, cool-down, yoga, and discussion. This group also receives the Treatment as Usual groups.
  Interventions: Behavioral: OT-led Exercise Group
- Treatment As Usual - OT Groups on Inpatient Psychiatry Unit (Placebo Comparator): An occupational therapist (OT) will begin daily educational session about the topic of choice for that day.
  Interventions: Behavioral: Treatment as Usual - OT Groups

INTERVENTIONS:
Behavioral: OT-led Exercise Group — Participants will complete pre-intervention self-report surveys about mood, anxiety, energy, self-esteem, and activity handed out by the research team. At this point, an occupational therapist (OT) will begin 10-minute educational session that describes the purpose of the exercise intervention and methods to remain safe during the intervention such as self-monitoring techniques. Following completion of the educational session, participants will complete a 30-minute exercise intervention under the guidance of the OT, which includes warm-up, high intensity interval training cardio, strength, kick boxing, cool-down, and yoga. Following completion of the exercise regimen, participants will participate in a 10-minute discussion and reflection with the OT and complete post-intervention self-report surveys. Participants in the intervention arm will also receive routine daily occupational therapy educational sessions received by the treatment as usual arm.
  Arms: OT-led Exercise Group on Inpatient Psychiatry Unit
Behavioral: Treatment as Usual - OT Groups — Participants will complete pre-session self-report surveys about mood, anxiety, energy, self-esteem, and activity handed out by the research team. At this point, an occupational therapist (OT) will begin daily educational session about the topic of choice for that day. Treatment groups are largely discussion-based and include the following topics: coping skills, self-esteem, sleep management, leisure, time management, life skills, decision making, and goal setting. Following completion of the educational session, participants will complete post-intervention self-report surveys.
  Arms: Treatment As Usual - OT Groups on Inpatient Psychiatry Unit

SUMMARY:
More research is needed to elucidate the impacts of physical activity interventions on short- and long-term activity and neuropsychiatric symptoms (NPS) in psychiatric inpatients and to support its advantageousness when compared to current standards of care. To investigate the impact of regular exercise on activity level, NPS, and sleep in an inpatient psychiatry unit, the investigators propose a placebo-controlled study with measures of activity, mood, anxiety, energy, and sleep as primary outcomes in 50 psychiatric inpatients at Johns Hopkins Hospital. Given the challenges of maintaining blinded assignment to treatment arm, the investigators will compare patients during two time periods (3 months each): the first is treatment as usual (TAU), the second adds exercise intervention (EXI).

DETAILED DESCRIPTION:
Growing evidence suggests that physical activity is associated with increased cognitive functioning and improved mental health. A recent meta-analysis demonstrated an inverse, dose-response association between physical activity and depression, particularly at lower activity volumes. Similarly, exercise has been shown to be associated with decreased anxiety, improved sleep, and reduced cognitive deficits in outpatient settings.

Despite the beneficial impacts of regular physical activity on mental health, physical activity is often low in psychiatric inpatient settings. Common barriers to exercise include lack of time and resources, limited staff knowledge, and competing treatment priorities. Organizational policy such as strict security procedures and restricted patient movement may also limit consistent integration of exercise into care. Finally, individuals with severe mental illness more commonly have sedentary lifestyles and may experience sedative side-effects of medication, which further limit ability to engage in physical activity.

There is limited literature on the impact of interventions aimed at increasing physical activity in psychiatric inpatient settings, however preliminary research suggests that these interventions may have positive short-term impacts on patients' mood and self-esteem. Investigators have found that over 90% of inpatients noted improved mood and body perception immediately following a structured exercise program. Moreover, there is evidence that psychiatric inpatients have a positive viewpoint of psychical activity intervention as part of psychiatric treatment and believe it will benefit the patients health. Given these findings, more research is needed to elucidate the impacts of physical activity interventions on short- and long-term activity and neuropsychiatric symptoms (NPS) in psychiatric inpatients and to support its advantages when compared to current standards of care.

Thus, to investigate the impact of regular exercise on activity level, NPS, and sleep in an inpatient psychiatry unit, the investigators propose a placebo-controlled study with measures of activity, mood, anxiety, energy, and sleep as primary outcomes in 60 psychiatric inpatients at Johns Hopkins Hospital. Half of the participants will be assigned to the exercise intervention (EXI) group, and the other half will be assigned to the treatment as usual (TAU) group. Group assignment will be made based on timing of study enrollment - the first 30 participants will be assigned to the TAU group, while the subsequent 30 participants will be assigned to the EXI group. Activity will be measured via actigraphy and self-report.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric inpatients admitted to the Johns Hopkins Bayview Acute Psychiatric Unit (APU)
* Aged 18 years or older
* Able to give informed consent and understand the tasks involved
* In the opinion of the unit attending, the patient is sufficiently psychologically or medically stable to safely participate in the exercise intervention
* Patients using mobility devices such as canes, walkers, and wheelchairs are eligible for inclusion as exercises can be completed in modifiable positions as needed.

Exclusion Criteria:

* Patients who do not speak English as their primary language.
* Patients with a history of physical or neurological conditions that interfere with study procedures.
* Patients demonstrating behavior that would be a safety concern if placed in a group at the discretion of occupational therapy, the medical team, or the nursing team.
* A patient can be excluded if in the opinion of the treatment team on the unit, participation in the study would have a negative impact on the patient's mental health or treatment plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in depression using Patient Health Questionnaire-9 | baseline, time of discharge up to 6 months
  Patient Health Questionnaire-9, range 0-27, lower score better outcome
Change in anxiety using Generalized Anxiety Disorder-7 | baseline, time of discharge up to 6 months
  Generalized Anxiety Disorder-7, range 0-21, lower score better outcome
Change in sleep using Pittsburgh Sleep Quality Index | baseline, time of discharge up to 6 months
  Pittsburgh Sleep Quality Index, range 0-21, lower score better outcome

SECONDARY OUTCOMES:
Length of Stay | time of discharge up to 6 months
  Length of stay will be collected via retrospective patient chart review or from patient care team upon discharge

CONTACTS AND LOCATIONS:
Overall Officials: Matthew E Peters, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States